CLINICAL TRIAL: NCT01696656
Title: Prescription Pattern of Adjuvant Drugs and Vitamins in Patients Undergoing Long-term Home Nutritional Support for Intestinal Insufficiency
Status: Completed | Type: Observational
Sponsor: University of Sao Paulo (Other)
Responsible Party: Principal Investigator, Joel Faintuch, Associate Professor, Department of Gastroenterology, Sao Paulo University Medical School, University of Sao Paulo
Other Study IDs: Gutadjuvant1; 0540/11 (Other: USaoPaulo)
Record Dates: First submitted 2012-09-27; First posted 2012-10-01 (Estimated); Last update posted 2012-10-01 (Estimated); Status verified 2012-09

CONDITIONS: Intestinal Insufficiency; Short Bowel Syndrome
Keywords: Gastrointestinal drugs; Antibiotics; Vitamins; Minerals; Intestinal insufficiency; Short Bowel syndrome; Adjuvant therapy; Antacids; Gastrointestinal motility modifiers; Micronutrients
MeSH Terms: conditions — Short Bowel Syndrome | interventions — Gastrointestinal Agents; Anti-Bacterial Agents; Vitamins; Minerals

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Intestinal insufficiency: Patients with variable categories of major intestinal resection due to benign diseases,suffering from intestinal insufficiency and maintained with home nutritional support. Only clinically stable and nonhospitalized subjects will be recruited.
  Interventions: Drug: Drug prescription pattern

INTERVENTIONS:
Drug: Drug prescription pattern — Type, dosage, administration route and frequency of prescription of all adjuvant pharmacologic agents will be transcribed from hospital records
  Other Names: Gastrointestinal drugs; Antibiotics; Vitamins; Minerals; General drugs

SUMMARY:
Intestinal insufficiency due to short bowel syndrome is a chronic, disabling condition with significant morbidity and mortality.Standard care includes home parenteral/enteral nutrition as well as intestinal transplantation, however multiple drugs, vitamins, antibiotics and symptom-relieving agents may be required. Prescriptional pattern of these drugs will be analyzed in a clinical cohort.

DETAILED DESCRIPTION:
Intestinal insufficiency due to short bowel syndrome is a chronic, disabling condition with significant morbidity and mortality.Standard care includes home parenteral/enteral nutrition as well as intestinal transplantation, however multiple drugs, vitamins, antibiotics and symptom-relieving agents may be required. Little attention has been given to the indications and dosage schedules of such drugs, many of which are employed as off-label prescriptions because of lack of official guidelines.

Prescriptional patterns of these drugs will be analyzed in a clinical cohort of home parenteral/enteral nutrition patients, registered at the outpatient service of Hospital das Clinicas, Sao Paulo, Brazil.

ELIGIBILITY:
Inclusion Criteria: Home nutritional support longer than 12 months,full records and return visits available at the hospital system.

-

Exclusion Criteria: Critical illness, death, discontinuation of nutritional therapy, registered for intestinal transplantation, additional gastrointestinal operations for short bowel syndrome (valves, lengthening) or for other conditions (gallbladder disease, intestinal obstruction, necrosis, infection).

-

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adults with short bowel syndrome secondary to trauma, Crohn´s disease, mesenteric thrombosis, radiation enteritis and other conditions, suffering from intestinal insufficiency and undergoing home-parenteral or enteral nutrition.
Sampling Method: Non-Probability Sample
Enrollment: 37 (Actual)
Dates: Start 2012-09; Primary Completion 2012-09 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Major gastrointestinal adjuvant prescription | Last 12 months
  The most prescribed adjuvant agent for alleviation of gastrointestinal troubles such as diarrhea, malabsorption or gastric hypersecretion.

SECONDARY OUTCOMES:
Major antibiotic adjuvant prescription | Last 12 months
  Principal antibiotic employed for suspected or actual bacterial overgrowth associated with diarrhea, malabsorption or systemic aberrations.

OTHER OUTCOMES:
Main vitamin/mineral adjuvant prescription | Last 12 months
  Vitamin, mineral or other micronutrient required for correction of nutrition deficiency, not available or poorly absorbed via current parenteral/enteral nutrition regimen

CONTACTS AND LOCATIONS:
Overall Officials: Bruna Z Godoy, RPh, Principal Investigator — University of Sao Paulo
Locations (1):
- Hospital das Clinicas- Central Institute ICHC- 9th Floor Rm 9077, São Paulo, São Paulo, Brazil

REFERENCES:
- [Background] Tilg H. Short bowel syndrome: searching for the proper diet. Eur J Gastroenterol Hepatol. 2008 Nov;20(11):1061-3. doi: 10.1097/MEG.0b013e3283040cc9. PMID 19047836
- [Background] Thompson JS, Rochling FA, Weseman RA, Mercer DF. Current management of short bowel syndrome. Curr Probl Surg. 2012 Feb;49(2):52-115. doi: 10.1067/j.cpsurg.2011.10.002. No abstract available. PMID 22244264
- [Background] Efsen E, Jeppesen PB. Modern treatment of adult short bowel syndrome patients. Minerva Gastroenterol Dietol. 2011 Dec;57(4):405-17. PMID 22105729